CLINICAL TRIAL: NCT07350304
Title: Comparison of Two OCT Device RNFL and GCIPL Measurements in Mild, Moderate, and Severe Glaucoma
Status: Completed | Type: Observational
Sponsor: Twin Cities Eye Consultants (Other)
Collaborators: Topcon Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: TCEC-001
Record Dates: First submitted 2025-12-29; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-12

CONDITIONS: Glaucoma
Keywords: Glaucoma; OCT; Optical Coherence Tomography
MeSH Terms: conditions — Glaucoma | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Derivation: The derivation cohort consisted of the first 72 eyes enrolled in the study. These participants had established glaucoma and were selected consecutively from a single clinical practice. Each eye underwent back-to-back OCT imaging using both the Topcon Maestro2 and Zeiss Cirrus 5000 devices during the same visit. Data from this cohort were used to develop statistical conversion models assessing agreement and potential equivalence in RNFL and GCIPL thickness measurements across platforms.
  Non-interventional imaging procedures were performed using standard manufacturer-recommended scan protocols. These included the Topcon Wide Scan, RNFL Cube, and Macular Cube protocols, as well as the Zeiss Optic Disc Cube 200×200 and Macular Cube 512×128 protocols. All scans were conducted by a single trained technician under controlled clinical conditions.
  Interventions: Diagnostic Test: Optical Coherence Tomography
- Validation: The validation cohort included the subsequent 69 eyes enrolled in the study, following the derivation cohort. Imaging procedures and clinical characteristics mirrored those of the derivation group. This cohort was used to test and validate the accuracy and reliability of the conversion models derived from the initial group.
  Subjects underwent the same non-invasive imaging protocols on both the Topcon Maestro2 and Zeiss Cirrus 5000 devices during a single clinic session. Scan protocols, technician, and environmental conditions were consistent with those of the derivation cohort to preserve standardization.
  Interventions: Diagnostic Test: Optical Coherence Tomography

INTERVENTIONS:
Diagnostic Test: Optical Coherence Tomography — Subjects underwent bilateral Optical Coherence Tomography (OCT) imaging using both the Topcon Maestro2 and Zeiss Cirrus 5000 devices during the same clinical session. Manufacturer-recommended protocols were used: Wide Scan, RNFL Cube, and Macular Cube (Topcon), and Optic Disc Cube 200×200 and Macular Cube 512×128 (Zeiss). Imaging was performed back-to-back using factory-default settings and standardized pupil dilation to assess cross-platform agreement and repeatability of RNFL and GCIPL thickness measurements in glaucomatous eyes.
  Other Names: OCT; Maestro2; Cirrus 5000

SUMMARY:
This research study was designed to evaluate how consistently two different imaging devices measure the thickness of retinal layers in patients with glaucoma. The two machines, the Topcon Maestro2 and the Zeiss Cirrus 5000, are commonly used in eye clinics to take high-resolution scans of the retina and optic nerve. These scans help doctors monitor glaucoma and detect disease progression.

The goal of this study was to compare the results from both machines when scanning the same patients, and to determine how closely their measurements align. Researchers also developed mathematical models that allow doctors to convert results from one machine to the other, which could help ensure consistency when a patient receives scans on different devices over time or at different clinics.

A total of 141 eyes from patients with varying levels of glaucoma severity were included in the study. Scans were performed using standard imaging protocols on both machines. Researchers analyzed the average thickness of two important retinal layers: the retinal nerve fiber layer (RNFL) and the ganglion cell-inner plexiform layer (GCIPL).

This study helps improve our understanding of how different imaging devices compare and provides tools for standardizing results across platforms. The findings may help eye care providers make more confident decisions when reviewing images from different machines, improving the care and monitoring of patients with glaucoma.

This was an investigator-initiated study sponsored by Twin Cities Eye Consultants with funding support from Topcon Healthcare. No new medications, treatments, or procedures were tested as part of this research. The study only involved non-invasive eye imaging scans that are already widely used in clinical practice.

DETAILED DESCRIPTION:
This investigator-initiated, cross-sectional study was designed to assess the level of agreement between optical coherence tomography (OCT) measurements captured by two commercially available imaging platforms: the Topcon Maestro2 and the Zeiss Cirrus 5000. These devices are widely used in the clinical management of glaucoma to quantify structural biomarkers such as retinal nerve fiber layer (RNFL) thickness and ganglion cell-inner plexiform layer (GCIPL) thickness.

The motivation behind this study stems from real-world variability in imaging hardware across clinical settings. Patients may undergo imaging on different machines due to equipment availability, clinic referral patterns, or evolving device infrastructure. As each device uses proprietary software algorithms and scan acquisition protocols, there can be small but clinically significant differences in reported measurements-even when scanning the same eye under similar conditions. Understanding this variability is critical for ensuring continuity of care and accuracy in longitudinal monitoring of glaucoma.

The study enrolled 141 eyes from patients with established glaucoma, screened from a single clinical practice. The first 72 eyes enrolled were designated as the derivation cohort, while the subsequent 69 eyes comprised the validation cohort. Each subject underwent back-to-back imaging on both devices during the same session using manufacturer-recommended scan protocols: the Topcon Wide Scan, RNFL Cube, and Macular Cube protocols; and the Zeiss Optic Disc Cube 200×200 and Macular Cube 512×128 protocols. All imaging was performed by a single, trained technician using factory-default acquisition settings and standard dilation (phenylephrine 2.5% and tropicamide 1%), with eye-tracking (FastTrac) enabled where available.

Average RNFL thickness and GCIPL thickness were extracted from each scan and compared between devices. Measurements were further analyzed by quadrant (RNFL) and sector (GCIPL) to evaluate regional agreement. Generalized linear models and Deming regression were used to evaluate the level of agreement and construct conversion equations between devices. Results were evaluated based on clinical thresholds of ±3 microns-a commonly accepted tolerance for scan-to-scan variability on a single device.

Repeatability of Topcon scans was also assessed using three consecutive scans on the same visit. Intra-device variability was analyzed using mean differences and 95% limits of agreement to determine reliability across protocols. Exploratory subgroup analyses were performed by glaucoma severity, gender, race/ethnicity, and visual acuity to explore potential drivers of scan variability or poor agreement.

The study found that while mean RNFL and GCIPL measurements from the two devices were highly correlated, statistically significant differences in average values were observed. This reinforces the importance of accounting for device-specific variability in both research and clinical practice. Derived conversion equations demonstrated strong performance in the validation cohort, particularly for global RNFL and GCIPL metrics. Sector-level agreement was more variable, particularly in the temporal RNFL and superotemporal GCIPL sectors, indicating that clinicians should use caution when interpreting regional values across platforms.

Importantly, scan repeatability on the Maestro2 was excellent, particularly for macular GCIPL metrics, highlighting its reliability for longitudinal monitoring. This supports the growing role of widefield and integrated OCT imaging in clinical glaucoma care.

The study was approved by Sterling IRB and conducted at Twin Cities Eye Consultants (Minnesota). It involved no investigational treatments or interventions beyond standard OCT imaging. Funding support was provided by Topcon Healthcare, which had no role in study design, data analysis, or manuscript preparation. Results from this study are intended to inform clinicians, researchers, and device manufacturers regarding the interoperability and clinical translation of OCT imaging biomarkers in glaucoma.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients at least 18 years of age
* A diagnosis of mild, moderate or severe glaucoma.
* Optic nerve appearance characteristic of glaucoma.
* < +/- 6D Spherical equivalent Refractive Error
* BCVA ≥ 20/40
* Previous Zeiss OCT RNFL with signal strength of ≥ 7/10
* The subject is able to understand the requirements of the study and provide written informed consent.
* Subject is willing to follow study instructions, agrees to comply with all study procedures and testing.

Exclusion Criteria:

* If pseudophakic, PCO must be ≤ trace
* If phakic, the cataract must be ≤ 1+
* No diagnosis of optic nerve disease other than glaucoma, and no macular disease.
* Current participation or participation in any drug or device clinical trial (which includes the fellow eye) within the past 30 calendar days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population consisted of adult patients aged 18 years or older with established or suspected glaucoma. Subjects were consecutively enrolled from a single tertiary ophthalmology practice in Minnesota. The final cohort included a range of glaucoma severity (mild, moderate, and severe) and was predominantly composed of White (59.6%) and female (59.6%) individuals. All participants underwent same-day, back-to-back OCT imaging on both the Topcon Maestro2 and Zeiss Cirrus 5000 systems.
Sampling Method: Non-Probability Sample
Enrollment: 141 (Actual)
Dates: Start 2024-10-28 (Actual); Primary Completion 2025-02-14 (Actual); Study Completion 2025-02-14 (Actual)

PRIMARY OUTCOMES:
Agreement Between Topcon Maestro2 and Zeiss Cirrus 5000 OCT Devices | Day of single study visit
  This primary outcome evaluates the cross-platform agreement of retinal nerve fiber layer (RNFL) and ganglion cell-inner plexiform layer (GCIPL) thickness measurements between the Topcon Maestro2 and Zeiss Cirrus 5000 devices in glaucoma and glaucoma-suspect eyes. The analysis will assess absolute differences, standard deviation, 95% limits of agreement, and proportion of eyes within a ±3 micron threshold for global and sectoral measurements.

SECONDARY OUTCOMES:
Repeatability of Topcon Maestro2 OCT Measurements | Day of single study visit
  Evaluate the test-retest repeatability of RNFL and GCIPL thickness measurements acquired with the Topcon Maestro2 Wide, RNFL Cube, and Macular Cube scan protocols. Repeatability will be assessed using standard deviation of repeated measures, coefficient of variation (CV), and intraclass correlation coefficients (ICC) when applicable.
Impact of Glaucoma Severity on Device Agreement | Day of single study visit
  Assess whether glaucoma severity (mild, moderate, or severe) influences agreement between RNFL and GCIPL thickness values measured by the Topcon Maestro2 and Zeiss Cirrus 5000. Stratified analyses will be conducted for both derivation and validation cohorts.
Cross-Device Agreement by Quadrant and Sectoral Analysis | Day of single study visit
  Evaluate device agreement on a quadrant-by-quadrant and sectoral basis for both RNFL and GCIPL layers. The analysis will include superior, inferior, nasal, and temporal quadrants for RNFL, and superotemporal, superonasal, inferotemporal, and inferonasal sectors for GCIPL.
Predictive Modeling to Convert Measurements Between Devices | Day of single study visit
  Develop linear regression models using the derivation cohort to predict Zeiss Cirrus RNFL and GCIPL values based on Topcon Maestro2 outputs. Validate model performance in a separate validation cohort within ±3 microns.

CONTACTS AND LOCATIONS:
Locations (1):
- Twin Cities Eye Consultants, Coon Rapids, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Tan O, Chopra V, Lu AT, Schuman JS, Ishikawa H, Wollstein G, Varma R, Huang D. Detection of macular ganglion cell loss in glaucoma by Fourier-domain optical coherence tomography. Ophthalmology. 2009 Dec;116(12):2305-14.e1-2. doi: 10.1016/j.ophtha.2009.05.025. Epub 2009 Sep 10. PMID 19744726
- [Background] Wong E, Yoshioka N, Kalloniatis M, Zangerl B. Cirrus HD-OCT short-term repeatability of clinical retinal nerve fiber layer measurements. Optom Vis Sci. 2015 Jan;92(1):83-8. doi: 10.1097/OPX.0000000000000452. PMID 25479451
- [Background] Kotowski J, Wollstein G, Folio LS, Ishikawa H, Schuman JS. Clinical use of OCT in assessing glaucoma progression. Ophthalmic Surg Lasers Imaging. 2011 Jul;42 Suppl(0):S6-S14. doi: 10.3928/15428877-20110627-01. PMID 21790113
- [Background] Vazirani J, Kaushik S, Pandav SS, Gupta P. Reproducibility of retinal nerve fiber layer measurements across the glaucoma spectrum using optical coherence tomography. Indian J Ophthalmol. 2015 Apr;63(4):300-5. doi: 10.4103/0301-4738.158064. PMID 26044467
- [Background] Mwanza JC, Oakley JD, Budenz DL, Anderson DR; Cirrus Optical Coherence Tomography Normative Database Study Group. Ability of cirrus HD-OCT optic nerve head parameters to discriminate normal from glaucomatous eyes. Ophthalmology. 2011 Feb;118(2):241-8.e1. doi: 10.1016/j.ophtha.2010.06.036. Epub 2010 Oct 28. PMID 20920824